CLINICAL TRIAL: NCT06855602
Title: A Single Arm Pilot Study of the Chinese Herbal Medicine Formula (S-2196) for the Female Stress Urinary Incontinence (SUI)
Brief Title: CHM for Female Stress Urinary Incontinence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Prof., Hong Kong Baptist University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/23-24/0483
Record Dates: First submitted 2024-11-29; First posted 2025-03-04 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-02

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: stress urinary incontinence; female
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Chinese herbal medicine decoction
  Interventions: Drug: Chinese herbal medicine formula (S-2196)

INTERVENTIONS:
Drug: Chinese herbal medicine formula (S-2196) — During the 2-week intervention, all participants are required to take 150ml of S-2196 decoction (a Chinese herbal medicine formula containing four herbs) twice per day

SUMMARY:
This single-arm, open-label pilot clinical trial will test the hypothesis that S-2196, a Chinese herbal medicine formula, will show efficacy and safety in alleviating the amount and frequency of urinary incontinence in female individuals with stress urinary incontinence. All participants (n=15) will receive 1 week of screening, 2 weeks of intervention, and 1 week of follow-up.

DETAILED DESCRIPTION:
Purpose of the Study: This clinical study aims to observe the efficacy and safety of treating stress urinary incontinence in females using the Chinese herbal medicine formula S-2196.

Study Design: Single-arm, open-label, pilot trial.

Target Population: Female patients aged 55 years and above who meet the clinical diagnostic criteria for SUI set by the International Consultation on Urological Diseases (ICUD); and with the amount of urinary leakage >10g in the 1-hour pad test; capable of understanding and using Chinese; and have signed the informed consent form.

Sample Size: This clinical trial is an exploratory pilot study with an estimated sample size of 15 participants.

Treatment Plan: Participants will take the Chinese herbal medicine formula decoction for two weeks, twice a day, 150 milliliters each time, after meals.

Primary Outcome:

1. Change in the amount of urinary leakage in the 1-hour standard pad test, compared to baseline (Time point: after 2 weeks of treatment);
2. Change in average daily frequency of urinary incontinence episode, compared to baseline (Time point: after 2 weeks of treatment)

Secondary Outcome: Change in the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) score, compared to baseline (Time point: after 2 weeks of treatment)

Safety Outcomes:

1. Any adverse reaction symptoms/adverse events occurring after the trial treatment.
2. General physical examination items (including heart rate, blood pressure, etc.)

Statistical Analysis: The database is constructed using REDCap, and all statistics are analyzed using SPSS version 23 statistical analysis software, to analyze the general conditions, demographic and other baseline characteristics, compliance, efficacy, and safety of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥55 years
* Meet the ICUD diagnostic criteria of stress urinary incontinence
* Measured urine leakage >10g in the 1-hour standard pad test
* Understand and can follow written and verbal instructions in Chinese
* Able to independently use and complete the electronic diary during the 1-week screening period
* The subject is informed and voluntarily signs the informed consent form

Exclusion Criteria:

* Patients with other types of urinary incontinence, such as neurogenic urinary incontinence, urge urinary incontinence, and overflow urinary incontinence.
* Subjects with the following urogenital system diseases (vesicoureteral reflux, detrusor instability, congenital urethral abnormalities, urinary tract infection or hematuria indicated by routine urinalysis or urine culture, urogenital fistula, urethral diverticulum, bladder stones, urinary system tumors, abnormal vaginal bleeding, pelvic malignant tumors, uterine prolapse grade II or above).
* History of SUI surgery or complex urethral surgery, including previous transvaginal tension-free mid-urethral sling, anterior wall prolapse repair, urethral injection therapy, etc.
* Previous pelvic radiotherapy, radical surgery for pelvic malignant tumors, and pelvic floor surgery.
* Currently receiving or needing to continue treatment related to urinary incontinence, including pelvic floor muscle training, physical therapy, pessary, and medication.
* If using medications that affect urination during the screening period (including but not limited to thiazolidinediones, sodium-glucose cotransporter 2 inhibitors, anticholinergics, alpha- and beta-adrenergic receptor antagonists, alpha- and beta-adrenergic receptor agonists, diuretic antihypertensive drugs, antihistamines, M receptor antagonists, calcium channel blockers, angiotensin-converting enzyme inhibitors, hormonal drugs, neurotransmitter drugs, intestinal flora regulating drugs, etc.), and unable to maintain a stable dose during the study period; or if considering using the above medications during the study period but not using them during the screening period.
* Presence of neurological disorders (including but not limited to central nervous system injury, motor neuron disease, neurodegenerative diseases), diabetes, connective tissue diseases, mental disorders, hypertension (defined as long-term monitored systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg), severe cardiovascular and cerebrovascular diseases, severe liver or kidney diseases.
* Combined with chronic cough diseases such as chronic obstructive pulmonary disease (COPD), gastrointestinal diseases affecting drug absorption, or other chronic diseases in an unstable state.
* History of adverse reactions to traditional Chinese medicine, or G6PD deficiency.
* Unable to complete exercises such as walking or climbing stairs.
* Deemed unsuitable for participation in this study by the researchers due to psychological or physical reasons.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
The change in the amount of urine leakage during the 1-hour standard pad test compared to the baseline (time point: the end of the 2nd week of treatment) | Baseline, week2
  The measurement of leakage volume follows the standardized 1-hour pad test protocol by the International Continence Society (ICS). The procedure includes the following steps: (1) Participants are required to void their bladder 2 hours before the test. (2) Upon start, participants will wear a pre-weighed pad and are instructed to drink 500 milliliters of water within 15 minutes. (3) Participants will walk for 30 minutes, including walking up and down one flight of stairs. (4) Participants will perform the following activities during the remaining time: sit down and stand up 10 times, cough vigorously 10 times, run in place for 1 minute, bend down to pick up an object from the floor 5 times, and wash hands under running water for 1 minute. (5)After completing these activities, the pad will be weighed again to calculate the leakage volume. 1g < leakage volume ≤ 10g is classified as mild; 10g < leakage volume ≤ 50g is classified as moderate; leakage volume > 50g is defined as severe.
The change in the average daily frequency of urinary incontinence episode compared to the baseline (time point: the end of the 2nd week of treatment). | Baseline, week 2
  The average daily frequency of urinary incontinence episodes (IEF) is calculated based on the number of incidences of urinary incontinence within a continuous 24-hour period, as recorded in the patient-reported electronic bladder diaries.

SECONDARY OUTCOMES:
The Change in International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) score compared to baseline (Time point: after 2 weeks of treatment) | Baseline, week 2
  The ICIQ-SF is a questionnaire strongly recommended by the International Continence Society (ICS) for assessing stress urinary incontinence (SUI). It includes three questions regarding the frequency of incontinence, the amount of leakage, and the impact on daily life. The total score ranges from 0 to 21, with lower scores indicating less severe SUI.

OTHER OUTCOMES:
Safety Outcome: adverse events | Baseline, week 2, week 3
  All adverse events occur from the beginning of the participant's enrollment to the end of the trial, regardless of whether there is a casual relationship with the received treatments. It will be assessed by the number of adverse events recorded in the patient-reported electronic diary.
Safety Outcome: Heart rate (beats per minute, bpm) | Baseline, week 2, week 3
  Heart rate will be assessed by a registered Chinese medicine practitioner at each visit to reflect general physical condition safety.
Safety Outcome: Systolic and Diastolic Blood Pressure (millimeters of mercury, mmHg)) | Baseline, Week 2, Week 3
  Systolic and diastolic blood pressure will be assessed by a registered Chinese medicine practitioner at each visit to monitor blood pressure-related safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Baptist University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided